CLINICAL TRIAL: NCT07308691
Title: Evaluating a Novel Rehabilitation Chatbot: A Pilot Randomized Controlled Trial for Distal Radius Fracture Recovery
Acronym: OT FDR CHATBOT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB-2025-568-5
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Fracture Distal Radius
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot with conventional rehabilitation (Experimental): Participants receive standard outpatient occupational therapy rehabilitation for conservatively treated distal radius fractures (2 sessions/week for 12 weeks, focusing on range of motion, strengthening, and functional tasks) plus the "Wrist Health" mHealth chatbot for home-based rehabilitation. The chatbot delivers personalized daily home exercises, educational content on fracture recovery, adherence reminders, real-time progress tracking, and Q&A support.
  Interventions: Device: Wrist Health chatbot
- Conventional Rehabilitation Only (Active Comparator): Participants receive standard outpatient occupational therapy rehabilitation for conservatively treated distal radius fractures (2 sessions/week for 12 weeks) plus a conventional paper-based home exercise program. This includes printed instructions for daily wrist range of motion, strengthening, and functional exercises, with weekly paper exercise logs for self-monitoring. No digital tools, reminders, or interactive features are provided.
  Interventions: Other: Conventional DRF rehabilitation

INTERVENTIONS:
Device: Wrist Health chatbot — This intervention combines generative AI conversational interface with therapist backend monitoring. It supplements (does not replace) 2x/week outpatient occupational therapy, focusing on conservative distal radius fracture.
  Arms: Chatbot with conventional rehabilitation
Other: Conventional DRF rehabilitation — standard outpatient occupational therapy rehabilitation for conservatively treated distal radius fractures (2 sessions/week for 12 weeks) plus a conventional paper-based home exercise program. This includes printed instructions for daily wrist range of motion, strengthening, and functional exercises, with weekly paper exercise logs for self-monitoring. No digital tools, reminders, or interactive features are provided.
  Arms: Conventional Rehabilitation Only

SUMMARY:
This study is a single-center pilot randomized controlled trial evaluating a rehabilitation chatbot, "Wrist Health," for elderly patients (60-90 years) recovering from conservatively treated distal radius fractures in Hong Kong. The trial compares conventional hospital-based rehabilitation plus a conventional home program with the same conventional rehabilitation supplemented by the chatbot, which delivers home exercises, education, reminders, and real-time usage tracking. Participants are randomized 1:1, followed for 12 weeks, and assessed at baseline, week 6, and week 12 using functional measures (range of motion, grip and pinch strength, PRWE), satisfaction, quality of life (EQ-5D-5L), adherence, feasibility metrics, and Technology Acceptance Model-based usability and acceptance outcomes.

Data will be analyzed primarily on an intention-to-treat basis using appropriate parametric or non-parametric tests for between-group comparisons and repeated-measures methods to examine change over time, with qualitative feedback analyzed thematically. The study has obtained/will obtain ethics approval from relevant institutional review boards, uses informed consent procedures, and applies robust data protection measures (password-protected systems, anonymization, locked physical storage, and secure destruction after the retention period). The findings are expected to provide preliminary evidence on clinical usability, feasibility, and effectiveness of the chatbot and to inform the design of a larger, definitive RCT and potential integration of digital rehabilitation tools into routine practice for elderly distal radius fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-90 years and literate (able to read Chinese).
* Diagnosis of distal radius fracture (confirmed radiologically).
* Completed conservative treatment (post injury approximately 6 weeks) and cleared for active rehabilitation.
* Ability to provide informed consent and comply with study procedures.
* Access to a compatible smartphone or tablet for chatbot use.

Exclusion Criteria:

* Illiterate or unable to read Chinese.

  * Cognitive impairment or inability to follow Cantonese instructions.
  * Complications such as complex regional pain syndrome or open fractures with significant soft tissue injury.
  * Bilateral wrist fractures or previous fracture of the unaffected wrist.
  * Concurrent participation in another clinical trial.
  * Significant comorbidities limiting participation in rehabilitation (e.g., severe neurological or psychiatric illness)

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
PRWE change from baseline to 12 weeks (functional recovery) | Primary time point: 12 weeks
  The PRWE is a 15-item validated patient-reported questionnaire assessing wrist pain (5 items) and function/disability in daily activities (10 items), scored 0-100 (higher scores indicate worse pain/function). Participants complete it at baseline (post-fracture stabilization), 6 weeks, and 12 weeks post-rehabilitation start. This captures clinically meaningful recovery in elderly distal radius fracture patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lun Yan Ngan, Master, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- FHSS, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
small sample sizes, re-identification concerns, and resource limitations for data preparation.

REFERENCES:
- [Background] Amorosa LF, Vitale MA, Brown S, Kaufmann RA. A functional outcomes survey of elderly patients who sustained distal radius fractures. Hand (N Y). 2011 Sep;6(3):260-7. doi: 10.1007/s11552-011-9327-7. Epub 2011 Mar 8. PMID 22942849